CLINICAL TRIAL: NCT00677417
Title: A Retrospective Study Investigating the Diagnostic Value of Hyperbilirubinaemia as a Predictive Factor for Appendiceal Perforation in Acute Appendicitis
Brief Title: Diagnostic Value of Hyperbilirubinaemia as a Predictive Factor for Appendiceal Perforation in Acute Appendicitis
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Dr., Ruhr University of Bochum
Other Study IDs: 001
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Perforated Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The values of laboratory examinations which are useful for the diagnoses of appendicitis are white blood cell count (WBC), C-reactive protein (CRP) and erythrocyte blood sedimentation rate (ESR). However up to date there is no laboratory marker for the pre-operative diagnosis of appendiceal perforation in acute appendicitis. Recently hyperbilirubinaemia has been associated with appendiceal perforation. Aim of this retrospective study is therefore to investigate if hyperbilirubinaemia has a diagnostic value for the pre-operative diagnosis of appendiceal perforation in patients with appendicitis.

DETAILED DESCRIPTION:
We identified 538 patients with histologically proved acute appendicitis who underwent laparoscopic or conventional appendicectomy between January, 2004 and December, 2007 in a surgical department of an academic teaching hospital. A retrospective multiple chart review of the medical records including laboratory values (bilirubin, CRP, white blood count) and histological results was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Appendicitis and a preoperative laboratory workup with Leukocytes, C-reactive Protein, Bilirubin and liver transaminases GOT and GPT

Exclusion Criteria:

* Alcoholism
* A history of viral hepatitis
* Gilbert's disease
* Dubin Johnson syndrome
* BRIC (benign recurrent intra-hepatic cholestasis) and other documented biliary
* Hemolytic or liver diseases associated with hyperbilirubinaemia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are appendectomied and who received preoperative Liver function test (bilirubin, liver transaminases GOT and GPT)
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benno Mann, PD Dr. med., Principal Investigator — Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum, Germany; Michael Sand, Dr. med., Principal Investigator — Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum, Germany

REFERENCES:
- [Result] Sand M, Bechara FG, Holland-Letz T, Sand D, Mehnert G, Mann B. Diagnostic value of hyperbilirubinemia as a predictive factor for appendiceal perforation in acute appendicitis. Am J Surg. 2009 Aug;198(2):193-8. doi: 10.1016/j.amjsurg.2008.08.026. Epub 2009 Mar 23. PMID 19306980